CLINICAL TRIAL: NCT05373134
Title: Efficacy and Safety of Pentoxifylline in Improving Oxygenation in Hepatopulmonary Syndrome: A Randomized Double-blind Placebo-controlled Trial
Brief Title: Efficacy and Safety of Pentoxifylline in Improving Oxygenation in Hepatopulmonary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-HPS-02
Record Dates: First submitted 2022-04-13; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Hepatopulmonary Syndrome
MeSH Terms: conditions — Hepatopulmonary Syndrome | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline (Experimental): 400mg OD x 1 week, 400mg BD x 1 week then increased to 400mg TDS and continued
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo will be given in a same manner as experimental drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — 400mg OD x 1 week, 400mg BD x 1 week then increased to 400mg TDS and continued
  Arms: Pentoxifylline
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The triad of liver disease, arterial hypoxia, and extensive pulmonary vascular dilatation is known as the hepatopulmonary syndrome (HPS). The prevalence of this syndrome ranges from 10% to 30% in people with chronic liver disease.

The exact cause of HPS is unknown. Previous research has shown that eicosanoids function as vasoconstrictors and cause an increase in the number of intravascular macrophage-like cells. Cirrhosis has been linked to increased NO generation in the lungs, which has been linked to intrapulmonary venous dilation. Increased pulmonary NO production is attributed to increased expression of pulmonary vascular endothelial NO synthase (eNOS) and inducible NO synthase.

Increased hepatic synthesis and release of low levels of endothelin 1 (ET-1) has been established in recent investigations to function as a trigger for increasing eNO levels. TNF (tumor necrosis factor) and ET-1 have both been linked to the onset of experimental HPS. Increased CO generation and heme oxygenase expression have been linked to the progression of HPS in recent investigations. HPS increases mortality in cirrhotic patients and may affect the frequency and severity of portal hypertension consequences.

To the best of our knowledge there have been only three pilot studies in humans which checked the effect of pentoxifylline in hepatopulmonary syndrome and they showed highly contrasting results. The outcome was also measured in a short interval. Investigator hypothesize that pentoxifylline would improve the oxygenation in patients with hepatopulmonary syndrome

DETAILED DESCRIPTION:
Hypothesis Investigator hypothesize that pentoxifylline in hepatopulmonary syndrome would improve oxygenation by inhibiting TNF alpha and thereby reducing macrophage, endothelium induced NO production compared to placebo

Aim To study efficacy of pentoxifylline in reducing AaPO2 in hepatopulmonary syndrome when compared to placebo

Methodology:

Study design: Prospective double-blind randomized placebo-controlled trial DATA and SPECIMEN collection Patient data, demographics, etiology of liver disease, PFT, abdominal radiological studies will be collected 6-minute walk test will be done at the baseline, 3 months, and 6 months Sampling for ABG will be performed with the subject seated while breathing room air at baseline and at the end of 3 and 6 months and A-aPO2 values will be calculated using Alveolar gas equation.

TNF alpha levels, vWF, ET-1, VEGFR-3, iNOS, eNOS and IL-1 β levels will be measured at baseline and after 3 and 6 months.

DLCO and exhaled NO will be measured at the baseline and at the end of 3 and 6 months Blinding The study drug and placebo will be administered in identical packaging and labelling to ensure that investigators and participants are blinded to study treatment. The study drug and placebo will be labelled with a unique label letter that will be used to allocate treatment to the patient, but the allocation will not be indicated to the investigators or participants. Except for the trial pharmacists and biostatistician, no member of the study team or their extended personnel will have access to the randomization method during the study's execution. The investigator will get the treatment assignment from trial pharmacists in the case of a medical emergency in which breaking the blind is necessary to give medical care to the participant.

DEFINITION - Hepatopulmonary syndrome will be defined by

1. Presence of liver disease and / or portal hypertension AND
2. Partial pressure of oxygen <80mm Hg or Alveolar-arterial oxygen gradient [P (A-a)O2 gradient ≥ 15mmHg (0r 20 mmHg for patients >65 years] AND
3. Documented Intrapulmonary Vascular Dilatation by saline contrast echocardiogram

Sample size: Assuming that the improvement in oxygenation in the pentoxifylline group is 50% and that in the control group it would be 1%, with an alpha error of 5% and power of 90% investigator need to enroll 38 cases in the study.

Further assuming a dropout rate of 5% investigator need to enroll 40 cases randomized into two groups, 20 each, by block randomization method taking a block size of 4.

STATISTICAL ANALYSIS: Continuous data- Student's t test

* Nonparametric analysis- Mann Whitney test
* Survival outcome By Kaplan-Meier method curve.
* For all tests, p≤ 0.05 will be considered statistically significant.
* Analysis will be performed using SPSS.
* The analysis will be done with intention to treat and per protocol analysis if applicable.

Stopping rule:

Development of serious adverse effects leading to withdrawal of the drug or death from any cause Adverse events It is defined as the new onset event that is considered as a part of intervention which otherwise may be absent in absence of such intervention or therapy. All adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* Evidence of portal hypertension
* Intrapulmonary vascular dilatation in the form of shunting diagnosed on contrast echocardiogram
* AaPO2 > 15mmHg on seated room air (ABG) if age <65years and >20mmHg if Age≥ 70 years

Exclusion Criteria:

* Child C cirrhosis with CTP > 10 or with refractory ascites
* Intrinsic significant cardiopulmonary disease

  1. PFT indicating severe obstructive ventilatory defect (FEV1/FVC < 70)
  2. Hepatic hydrothorax, Portopulmonary hypertension
  3. Moderate and severe left ventricular systolic dysfunction
  4. Inability to perform Pulmonary function test
  5. Intracardiac shunting
* Current use of exogenous nitrates
* Patients already on pentoxifylline
* Prior intolerance to pentoxifylline
* Very severe cases of HPS (A-aO2 gradient ≥ 15mm Hg, PO2 <50 mmHg)
* Active bacterial infections, active hepatic encephalopathy
* Known malignancy including HCC
* SBP on secondary prophylaxis
* CKD with creatinine clearance < 30
* Enrolled in other trials
* Has a liver transplant option

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-05 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in AaPO2 gradient by at least 5mmHg or to a value less than 15mm Hg at the end of 6 months from baseline | 6 months

SECONDARY OUTCOMES:
Change in grading of intrapulmonary shunting at the end of 3 month, from baseline as assessed by saline contrast echocardiography | 3 months
Change in grading of intrapulmonary shunting at the end of 6 month, from baseline as assessed by saline contrast echocardiography | 6 months
Change in DLCO (Diffusing Capacity of the lungs for Carbon Monoxide) at the end of 3 month from baseline | 3 month
Change in Forced expiratory volume 1 (FEV1) at the end of 3 month from baseline | 3 month
Change in FVC (Forced Vital Capacity) at the end of 3 month from baseline | 3 month
Change in FEV1/FVC ratio at the end of 3 month from baseline | 3 month
Change in 6-minute walk test at the end of 3 month from baseline | 3 month
Change in DLCO (Diffusing Capacity of the lungs for Carbon Monoxide) at the end of 6 month from baseline | 6 month
Change in Forced expiratory volume 1 (FEV1) at the end of 6 month from baseline | 6 month
Change in FVC (Forced Vital Capacity) at the end of 6 month from baseline | 6 month
Change in FEV1/FVC ratio at the end of 6 month from baseline | 6 month
Change in 6-minute walk test at the end of 6 month from baseline | 6 month
Change in seated oxygen saturation at 3 month from baseline | 3 month
Change in PaO2 at 3 month from baseline | 3 month
Change in seated oxygen saturation at 6 month from baseline | 6 month
Change in PaO2 at 6 month from baseline | 6 month
Change in inflammatory markers at the end of 3 month from baseline | 3 month
  TNF alpha levels, vWF, ET-1, IL-6, S-1-P levels
Change in inflammatory markers at the end of 6 month from baseline | 6 month
  TNF alpha levels, vWF, ET-1, IL-6, S-1-P levels at the end of 6 month from baseline
Change in inflammatory markers at the end of 3 month from baseline in a subset of patients wherever feasible | 3 month
  VEGFR-3, iNOS, eNOS and IL-1 β
Change in inflammatory markers at the end of 6 month from baseline in a subset of patients wherever feasible | 6 month
  VEGFR-3, iNOS, eNOS and IL-1 β
Change in DLCO fraction of exhaled NO after 3 month from baseline | 3 month
Change in DLCO fraction of exhaled NO after 6 month from baseline | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided